CLINICAL TRIAL: NCT00001091
Title: A Phase II Rolling Arm Master Protocol (PRAM) of Novel Antiretroviral Therapy in Stable Experienced HIV-Infected Children. PRAM-2: A Phase I/II Randomized, Multicenter Protocol Comparing Four Antiretroviral Regimens Containing Combinations of Protease Inhibitors, NRTIs and an NNRTI
Brief Title: Safety and Effectiveness of Four Anti-HIV Drug Combinations in HIV-Infected Children and Teens
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: ACTG 377; 11338 (Registry Identifier: DAIDS ES); PACTG 377
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2021-11-04 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections
Keywords: Drug Therapy, Combination; Nevirapine; Stavudine; HIV Protease Inhibitors; Ritonavir; Lamivudine; Nelfinavir; Reverse Transcriptase Inhibitors
MeSH Terms: conditions — HIV Infections | interventions — Ritonavir; Nelfinavir; Nevirapine; Lamivudine; Stavudine

INTERVENTIONS:
Drug: Ritonavir
Drug: Nelfinavir mesylate
Drug: Nevirapine
Drug: Lamivudine
Drug: Stavudine

SUMMARY:
The purpose of this study is to see if it is safe and effective to give HIV-infected children and teens 1 of 4 anti-HIV drug combinations.

Decreasing HIV levels in infected patients can slow down disease progression. Further study is needed to find out which drug combinations are most effective in doing this.

DETAILED DESCRIPTION:
For PRAM 2: Evidence suggests that as a consequence of antiviral therapy, decreases in plasma HIV-1 RNA are strongly associated with a delay in clinical progression. Therefore, the drug regimens proposed in this study are designed to result in a much larger sustained drop in plasma HIV-1 RNA and greater clinical benefit. Further intent of this study is to evaluate the virologic and therapeutic potential of novel combinations of antiretrovirals and to better define the pharmacokinetics and drug-drug interactions of therapies included in this regimen.

The Master PRAM schema is designed to allow new therapeutic arms to be studied as "rolling screens" through multiple generations of PRAMs. There is a common, "linking" regimen between any 2 sequential PRAM generations that will permit an indirect comparison of included therapies. (NOTE: Due to significant changes in study design between PRAM 1 and PRAM 2, there is no "linking" arm between them. The linkage will be reinstated from PRAM 2 and subsequent PRAM generations.) The therapeutic potential of the treatment arms is assessed by their ability to decrease HIV copy numbers as defined by plasma HIV-1 RNA copy number. Once accrual to a PRAM is complete, a new treatment comparison will open for accrual.

For PRAM 2: This study will compare the following 4 treatment arms:

Arm A - stavudine (d4T)/nevirapine/ritonavir Arm B - d4T/lamivudine (3TC)/nelfinavir Arm C - d4T/nevirapine/nelfinavir Arm D - d4T/3TC/nevirapine/nelfinavir. Prior to randomization to 1 of the PRAM 2 treatment arms, patients are stratified based on their CD4% (less than 25% and greater than or equal to 25%) and by age (less than 24 months and greater than or equal to 24 months). The first 35 subjects/treatment arm are evaluated with special immunologic studies including lymphoproliferative assays and extended panel immunophenotyping. There is an interim analysis after all patients have completed 12 weeks of treatment. Patients are treated for 48 weeks. [AS PER AMENDMENT 6/11/99: The study has been extended for an additional 48 weeks (96 weeks total) to permit long-term follow-up of clinically stable, HIV-infected children.]

ELIGIBILITY:
Inclusion Criteria

Patients may be eligible for this study if they:

* Are HIV-positive.
* Have received the same continuous anti-HIV treatment for the past 16 weeks (missing no more than 6 weeks of treatment total during those 16 weeks).
* Are between 4 months and 17 years old (consent of parent or guardian required).

Exclusion Criteria

Patients will not be eligible if they:

* Have certain serious conditions such as cancer, an opportunistic (AIDS-related) infection, or other serious infection.
* Have ever taken any of the study drugs or any protease inhibitor.
* Are currently taking any anti-HIV drugs.
* Have taken an investigational drug within 14 days of entry into the study. (Co-enrollment in ACTG 219, ACTG 220 and certain ACTG opportunistic infection studies is allowed.)
* Are taking certain other drugs.
* Are pregnant.

Ages: 4 Months to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 200
Dates: Study Completion 2000-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Wiznia, Study Chair; George Johnson, Study Chair; Paul Krogstad, Study Chair
Locations (55):
- United States (53):
  - Univ of Alabama at Birmingham - Pediatric, Birmingham, Alabama
  - UCSD Med Ctr / Pediatrics / Clinical Sciences, La Jolla, California
  - Long Beach Memorial (Pediatric), Long Beach, California
  - Children's Hosp of Los Angeles/UCLA Med Ctr, Los Angeles, California
  - Los Angeles County - USC Med Ctr, Los Angeles, California
  - UCLA Med Ctr / Pediatric, Los Angeles, California
  - Harbor - UCLA Med Ctr / UCLA School of Medicine, Los Angeles, California
  - Children's Hosp of Oakland, Oakland, California
  - UCSF / Moffitt Hosp - Pediatric, San Francisco, California
  - Connecticut Children's Med Ctr - Pediatric, Hartford, Connecticut
  - Yale Univ Med School, New Haven, Connecticut
  - Children's Hosp of Washington DC, Washington D.C., District of Columbia
  - Washington Hosp Ctr, Washington D.C., District of Columbia
  - Howard Univ Hosp, Washington D.C., District of Columbia
  - North Broward Hosp District, Fort Lauderdale, Florida
  - Univ of Florida Gainesville, Gainesville, Florida
  - Univ of Florida Health Science Ctr / Pediatrics, Jacksonville, Florida
  - Palm Beach County Health Dept, Riviera Beach, Florida
  - Emory Univ Hosp / Pediatrics, Atlanta, Georgia
  - Med College of Georgia, Augusta, Georgia
  - Cook County Hosp, Chicago, Illinois
  - Univ of Illinois College of Medicine / Pediatrics, Chicago, Illinois
  - Chicago Children's Memorial Hosp, Chicago, Illinois
  - Univ of Chicago Children's Hosp, Chicago, Illinois
  - Tulane Univ / Charity Hosp of New Orleans, New Orleans, Louisiana
  - Univ of Maryland at Baltimore / Univ Med Ctr, Baltimore, Maryland
  - Johns Hopkins Hosp - Pediatric, Baltimore, Maryland
  - Baystate Med Ctr of Springfield, Springfield, Massachusetts
  - Univ of Massachusetts Med School, Worcester, Massachusetts
  - Univ of Mississippi Med Ctr, Jackson, Mississippi
  - UMDNJ - Robert Wood Johnson Med School / Pediatrics, New Brunswick, New Jersey
  - Saint Joseph's Hosp and Med Ctr/UMDNJ - New Jersey Med Schl, Newark, New Jersey
  - King's County Hosp Ctr / Pediatrics, Brooklyn, New York
  - SUNY - Brooklyn, Brooklyn, New York
  - North Shore Univ Hosp, Great Neck, New York
  - Schneider Children's Hosp, New Hyde Park, New York
  - Bellevue Hosp / New York Univ Med Ctr, New York, New York
  - Cornell Univ Med College, New York, New York
  - Metropolitan Hosp Ctr, New York, New York
  - Columbia Presbyterian Med Ctr, New York, New York
  - Incarnation Children's Ctr / Columbia Presbyterian Med Ctr, New York, New York
  - Harlem Hosp Ctr, New York, New York
  - Univ of Rochester Med Ctr, Rochester, New York
  - State Univ of New York at Stony Brook, Stony Brook, New York
  - Bronx Lebanon Hosp Ctr, The Bronx, New York
  - Bronx Municipal Hosp Ctr / Bronx Lebanon Hosp Ctr, The Bronx, New York
  - Bronx Municipal Hosp Ctr/Jacobi Med Ctr, The Bronx, New York
  - Children's Hosp of Philadelphia, Philadelphia, Pennsylvania
  - Saint Christopher's Hosp for Children, Philadelphia, Pennsylvania
  - Med Univ of South Carolina, Charleston, South Carolina
  - Vanderbilt Univ Med Ctr, Nashville, Tennessee
  - Children's Hosp of the King's Daughters, Norfolk, Virginia
  - Children's Hospital & Medical Center / Seattle ACTU, Seattle, Washington
- Puerto Rico (2):
  - Ramon Ruiz Arnau Univ Hosp / Pediatrics, Bayamón
  - San Juan City Hosp, San Juan

REFERENCES:
- [Background] Cunningham S, Ank B, Lewis D, Lu W, Wantman M, Dileanis JA, Jackson JB, Palumbo P, Krogstad P, Eshleman SH. Performance of the applied biosystems ViroSeq human immunodeficiency virus type 1 (HIV-1) genotyping system for sequence-based analysis of HIV-1 in pediatric plasma samples. J Clin Microbiol. 2001 Apr;39(4):1254-7. doi: 10.1128/JCM.39.4.1254-1257.2001. PMID 11283037
- [Result] Eshleman SH, Krogstad P, Jackson JB, Lee S, Wang YG, Wei LJ, Cunningham S, Wantman M, Lindquist C, Nachman S, Palumbo P. Analysis of HIV-1 drug resistance in a randomized, controlled trial of a combination of nucleoside analog reverse transcriptase (RT) inhibitors plus nevirapine (NVP), nelfinavir (NFV), or ritonavir (RTV) in stable antiretroviral therapy-experienced HIV-infected children. 8th Conf Retro and Opportun Infect. 2001 Feb 4-8 (abstract no 468)
- [Result] Eshleman SH, Krogstad P, Jackson JB, Wang YG, Lee S, Wei LJ, Cunningham S, Wantman M, Wiznia A, Johnson G, Nachman S, Palumbo P. Analysis of human immunodeficiency virus type 1 drug resistance in children receiving nucleoside analogue reverse-transcriptase inhibitors plus nevirapine, nelfinavir, or ritonavir (Pediatric AIDS Clinical Trials Group 377). J Infect Dis. 2001 Jun 15;183(12):1732-8. doi: 10.1086/320728. Epub 2001 May 16. PMID 11372025
- [Result] Krogstad P, Lee S, Johnson G, Stanley K, McNamara J, Moye J, Jackson JB, Aguayo R, Dieudonne A, Khoury M, Mendez H, Nachman S, Wiznia A; Pediatric AIDS Clinical Trials Group 377 Study Team. Nucleoside-analogue reverse-transcriptase inhibitors plus nevirapine, nelfinavir, or ritonavir for pretreated children infected with human immunodeficiency virus type 1. Clin Infect Dis. 2002 Apr 1;34(7):991-1001. doi: 10.1086/338814. Epub 2002 Feb 27. PMID 11880966
- [Result] Van Dyke RB, Lee S, Johnson GM, Wiznia A, Mohan K, Stanley K, Morse EV, Krogstad PA, Nachman S; Pediatric AIDS Clinical Trials Group Adherence Subcommittee Pediatric AIDS Clinical Trials Group 377 Study Team. Reported adherence as a determinant of response to highly active antiretroviral therapy in children who have human immunodeficiency virus infection. Pediatrics. 2002 Apr;109(4):e61. doi: 10.1542/peds.109.4.e61. PMID 11927734
- [Result] Wiznia A, Stanley K, Krogstad P, Johnson G, Lee S, McNamara J, Moye J, Jackson JB, Mendez H, Aguayo R, Dieudonne A, Kovacs A, Bamji M, Abrams E, Rana S, Sever J, Nachman S. Combination nucleoside analog reverse transcriptase inhibitor(s) plus nevirapine, nelfinavir, or ritonavir in stable antiretroviral therapy-experienced HIV-infected children: week 24 results of a randomized controlled trial--PACTG 377. Pediatric AIDS Clinical Trials Group 377 Study Team. AIDS Res Hum Retroviruses. 2000 Aug 10;16(12):1113-21. doi: 10.1089/088922200414956. PMID 10954886
- [Result] Jeremy RJ, Kim S, Nozyce M, Nachman S, McIntosh K, Pelton SI, Yogev R, Wiznia A, Johnson GM, Krogstad P, Stanley K; Pediatric AIDS Clinical Trials Group (PACTG) 338 & 377 Study Teams. Neuropsychological functioning and viral load in stable antiretroviral therapy-experienced HIV-infected children. Pediatrics. 2005 Feb;115(2):380-7. doi: 10.1542/peds.2004-1108. PMID 15687448
- [Result] Rosenblatt HM, Song LY, Nachman SA, Stanley KE, Krogstad PA, Johnson GM, Wiznia AA; Pediatric Aids Clinical Trials Group 377 Study Team. Tetanus immunity after diphtheria, tetanus toxoids, and acellular pertussis vaccination in children with clinically stable HIV infection. J Allergy Clin Immunol. 2005 Sep;116(3):698-703. doi: 10.1016/j.jaci.2005.05.016. PMID 16159645
- [Result] Saitoh A, Sarles E, Capparelli E, Aweeka F, Kovacs A, Burchett SK, Wiznia A, Nachman S, Fenton T, Spector SA. CYP2B6 genetic variants are associated with nevirapine pharmacokinetics and clinical response in HIV-1-infected children. AIDS. 2007 Oct 18;21(16):2191-9. doi: 10.1097/QAD.0b013e3282ef9695. PMID 18090046